CLINICAL TRIAL: NCT03938233
Title: A Scalable Solution for Delivery of Diabetes Self-Management Education in Thailand
Brief Title: Diabetes Self Management Education Programme in Thailand
Acronym: DSMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Medical Research Council (Other Government); Chiang Mai University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1
Record Dates: First submitted 2019-04-24; First posted 2019-05-06 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Self-management; Structured Education; Thailand; Peer Led
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Cluster randomised control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DSME program delivered by community health volunteers (Active Comparator): Randomisation will happen in 21 primary care units to offer DSME delivered by lay health workers to those newly diagnosed with diabetes and those having difficulties with self-managing their diabetes.
  Interventions: Behavioral: A low-cost DSME program and scalable delivery model for roll-out within the Thai primary care system
- DSME program delivered by nurses (Active Comparator): Randomisation will happen in 21 primary care units to offer DSME delivered by nurses (for comparative effectiveness) to those newly diagnosed with diabetes and those having difficulties with self-managing their diabetes.
  Interventions: Behavioral: A low-cost DSME program and scalable delivery model for roll-out within the Thai primary care system
- Usual care(no DSME program) (No Intervention): Randomisation will happen in 21 primary care units where no DSME will be offered to those newly diagnosed with diabetes and/or those having difficulties with self-managing their diabetes.These patients will continue with usual care and will be assessed as the control group.

INTERVENTIONS:
Behavioral: A low-cost DSME program and scalable delivery model for roll-out within the Thai primary care system — The intervention will be based on behaviour-change and social support theories, delivered in monthly group meetings by lay health workers or nurses, and aided by a suite of short films to introduce key topics and stimulate discussion.
  Arms: DSME program delivered by community health volunteers; DSME program delivered by nurses

SUMMARY:
Type 2 diabetes is amongst the foremost challenges facing policy makers in Thailand, accounting for considerable death, disability and healthcare expenditure. Under Thailand's strong primary health system, medical management of diabetes is widely available. However, control of blood glucose and other cardiovascular disease risk factors, and regular screening for early detection of complications remain low due to a lack of services for education and counselling to support behavioural changes necessary for good self-management of the condition. A substantial literature documents the effectiveness of Diabetes Self-Management Education (DSME) programs for improving diabetes outcomes, although little high-quality data are available in Thailand, and traditional delivery models (health-professional led one-to-one or small-group sessions) are unlikely to be scalable in Thailand given current human resource and budgetary constraints. Thus, a low-cost DSME program will be developed with a scalable delivery model for roll-out within the Thai primary care system. The intervention will be based on behaviour-change and social support theories, delivered in monthly group meetings by lay health workers or nurses, and aided by a suite of short films to introduce key topics and stimulate discussion. 21 primary care units will be randomised to offer to those with diabetes diagnosed within the first three years. DSME will be delivered by lay health workers, nurses (for comparative effectiveness), or usual care. After 12 months, glycaemic control and cardiovascular risk scores will be compared between the three arms. Cost-effectiveness will be assessed, also process and policy evaluations to produce best-buy recommendations for the Thai Ministry of Public Health.

DETAILED DESCRIPTION:
The health and economic consequences of Type 2 diabetes mellitus are largely attributable to its complications, which can be prevented or delayed by good disease control, achieved through medical care and self-management. Diabetes Self- Management Education (DSME) programs are effective and cost-effective, and part of standard care in high-income countries, but are unavailable in Thai healthcare system, despite universal coverage of medical aspects of diabetes care. Negative perceptions of educational programs, sustained by a lack of high-quality local data, and concerns about burden on existing staff time and costs are thought to be responsible.

Given the focus on community-based education for chronic diseases in recent primary healthcare reforms, it is timely to scale-up DSME in Thailand, if an affordable model of delivery for a locally-tailored intervention can be found. The aim is to work in close collaboration with the Thai Ministry of Public Health to develop, pilot and evaluate a peer-based DSME program and delivery model. A final list of policy recommendations for optimal integration into the Thai healthcare system will be produced.

The aim is to identify a scalable model for delivery of DSME across Thailand.

Specific project objectives are:

1. To design a prototype of the DSME intervention
2. To refine the intervention prototype and trial design
3. To evaluate the effectiveness and cost-effectiveness of the intervention under two alternative modes of delivery (nurse-led and peer-led)
4. To identify the 'best buy' model for scale-up of DSME delivery in the Thai health system.

The primary hypothesis is that either model of DSME delivery will be effective and cost-effective, but the peer-led model will be a more scalable option for the Thai health system.

The two key research gaps in scientific literature that will be addressed are:

1. Clinical and cost-effectiveness of DSME programs in low- and middle-income countries, specifically Thailand
2. Role of peer programs in supporting complex behaviour change generally, and its implementation in low- and middle-income settings specifically.

The main expected outcomes are:

1. Development of a fully worked-up rapidly scalable model for DSME delivery in Thailand;
2. Capacity building of emerging Thai researchers and practitioners (nurses, village health volunteers) in the science and delivery of complex behavioural interventions, which could be expanded to other chronic conditions;
3. Long-term collaborative research links between UK and Thai researchers.

ELIGIBILITY:
Inclusion Criteria:

* People aged over 18 years with a new referral for type-2 diabetes management at the 15 hospitals
* People aged over 18 years with difficulties managing type-2 diabetes up to three years of diagnosis at the 15 hospitals
* Willingness to attend educational group meetings
* Available for 12-month follow-up

Exclusion Criteria:

* Advanced diabetes complications such as receiving dialysis, registered blind, above ankle amputations.
* Co-morbid learning difficulties, dementia or severe mental illness
* Lacking the capacity to consent
* Those aged under 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 693 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c levels (HbA1c) | 12 months
  HbA1c will measures the average blood glucose (sugar) levels months
Total cardiovascular risk | 12 months
  The cardiovascular risk will be estimated by Systemic Coronary Risk Evaluation. (SCORE) model. This is a range from 120 to 180 measuring systolic blood pressure (mmHq).

SECONDARY OUTCOMES:
EQ-5D | 12 months
  Quality of Life measure that will also assess cost-effectiveness. Includes five quality of life question on mobility, self-care, usual activity, pain, anxiety / depression and a scale of 0 to 100 on how the person is feeling on that day.
  Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The respondent is asked to indicate his/her health state by ticking in the box against the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number expressing the level selected for that dimension. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.
Hospital Anxiety and Depression scale (HADS) | 12 months
  HADS measures depression and anxiety which will address psychological change. Scale is from 0 to 3.
  Scale defined as:
  Definitely 0 Usually 1 Sometimes 2 Not often 3 Not at all Total score of 21.
  Scoring:
  Total score:
  0-7 = Normal 8-10 = Borderline abnormal (borderline case) 11-21 = Abnormal (case)
Perceived Stress Questionnaire (PSQ) | 12 months
  PSQ will assess stress and ability to self-management. 30 questions on how the person is feeling with a scale from 1 to 4.
  0 = Never 1 = Almost Never 2 = Sometimes 3 = Fairly Often 4 = Very Often Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Summary of Diabetes Self-Care Activities Assessment (SDSCA) | 12 months
  Diabetes self-care activities questionnaire focuses on general diet, diabetes-specific diet, physical activity, blood-glucose testing, foot care, and smoking. With a scale of 0 to 7 with no cut of points. Higher score indicate higher self care activities.
International Physical Activity Questionnaire | 12 months
  The assessment of physical activity comprises a set of 4 questionnaires. Long (5 activity domains asked independently) and short (4 generic items) versions.There are two forms of output from scoring the IPAQ. Results can be reported in categories (low activity levels, moderate activity levels or high activity levels) or as a continuous variable (MET minutes a week). MET minutes represent the amount of energy expended carrying out physical activity.
  Expressed as MET-min per week:
  MET level x minutes of activity x events per week
  Sample Calculation:
  MET levels MET-min/week for 30 min episodes, 5 times/week Walking = 3.3 METs 3.3*30*5 = 495 MET-min/week Moderate Intensity = 4.0 METs 4.0*30*5 = 600 MET-min/week Vigorous Intensity = 8.0 METs 8.0*30*5 = 1,200 MET-min/week
  ___________________________ TOTAL = 2,295 MET-min/week Total MET-min/week = (Walk METs*min*days) + (Mod METs*min*days) + Vig METs*min*days)
Body mass index (BMI) | 12 months
  Height and weight (used to derive BMI)

OTHER OUTCOMES:
Smoking | 12 months
  Assessing the number of cigarettes smoked through four set questions. Do you currently use tobacco? 0 1 Yes, on a regular basis Number per day: ____________ 02 Yes, but only once in a while 03 Not anymore, I quit 04 No, I have never used tobacco

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Kinra, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made upon reasonable request

REFERENCES:
- [Derived] Papachristou Nadal I, Aramrat C, Jiraporncharoen W, Pinyopornpanish K, Wiwatkunupakarn N, Quansri O, Rerkasem K, Srivanichakorn S, Techakehakij W, Wichit N, Pateekhum C, Birk N, Ngetich E, Khunti K, Hanson K, Kinra S, Angkurawaranon C. Process evaluation protocol of a cluster randomised trial for a scalable solution for delivery of Diabetes Self-Management Education in Thailand (DSME-T). BMJ Open. 2021 Dec 9;11(12):e056141. doi: 10.1136/bmjopen-2021-056141. PMID 34887283
- [Derived] Angkurawaranon C, Papachristou Nadal I, Mallinson PAC, Pinyopornpanish K, Quansri O, Rerkasem K, Srivanichakorn S, Techakehakij W, Wichit N, Pateekhum C, Hashmi AH, Hanson K, Khunti K, Kinra S. Scalable solution for delivery of diabetes self-management education in Thailand (DSME-T): a cluster randomised trial study protocol. BMJ Open. 2020 Oct 5;10(10):e036963. doi: 10.1136/bmjopen-2020-036963. PMID 33020090

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03938233/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03938233/ICF_001.pdf